CLINICAL TRIAL: NCT01065181
Title: Shoulder Posterior Capsular Contracture in Youth Baseball Players: It Can be Improved by Stretching
Brief Title: Youth Throwers Respond to Stretching
Acronym: Safethrow
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Metzger, Charles, M.D. (Individual)
Responsible Party: Principal Investigator, Charles Metzger, M.D., Associate Program Director, Metzger, Charles, M.D.
Other Study IDs: Safethrow01
Record Dates: First submitted 2010-02-06; First posted 2010-02-09 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Shoulder Posterior Capsular Contracture
Keywords: shoulder; posterior inferior glenohumeral ligament; posterior capsule; capsular contracture; baseball; throwing injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to document the rates of youth baseball player demographics, incidence of arm pain, usage of different pitch types, and degree of internal rotation contracture in the throwing versus the non-throwing shoulder. We followed a subgroup of players for a year to see if a particular stretch would help reduce the internal rotation contracture.

DETAILED DESCRIPTION:
Introduction: Overhead throwing can cause contracture of the shoulder posterior-inferior glenohumeral ligament which can lead to injuries such as superior labral tears. We show that instruction on stretching can favorably alter progression of posterior contractures.

Methods: 1261 male baseball players ages 7-15 completed a questionnaire and shoulder examinations. Measurements of rotation of both shoulders were made with the subjects in the supine position with the scapula stabilized. Glenohumeral internal rotation deficit (GIRD) was calculated. Pitch type and player position, among other variables, were recorded. The prospective cohort was 175 players who were examined twice a year apart. Players with excessive GIRD (exGIRD) were given stretching instruction, and the control group was those without exGIRD who were not given instruction. Change in GIRD as a result of this intervention was documented.

ELIGIBILITY:
Inclusion Criteria:

* male
* baseball player
* ages 8 to 15

Exclusion Criteria:

* female (suspected hormonal/gender influences on capsular elasticity)
* prior throwing arm surgery

Ages: 8 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1261 male baseball players ages 8 to 15
Sampling Method: Non-Probability Sample
Enrollment: 1261 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Degree of decrease in internal rotation contracture of the shoulder | One year
  GIRD is the Glenohumeral Internal Rotation Deficit. It is the difference in the internal rotation of the throwing shoulder compared to the non-throwing shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Metzger, MD, Principal Investigator — Memorial Hermann Health System

REFERENCES:
- [Background] Lyman S, Fleisig GS. Baseball injuries. Med Sport Sci. 2005;49:9-30. doi: 10.1159/000085340. PMID 16247260
- [Background] Kerut EK, Kerut DG, Fleisig GS, Andrews JR. Prevention of arm injury in youth baseball pitchers. J La State Med Soc. 2008 Mar-Apr;160(2):95-8. PMID 18681352
- [Result] Awan R, Smith J, Boon AJ. Measuring shoulder internal rotation range of motion: a comparison of 3 techniques. Arch Phys Med Rehabil. 2002 Sep;83(9):1229-34. doi: 10.1053/apmr.2002.34815. PMID 12235602
- [Result] Lyman S, Fleisig GS, Waterbor JW, Funkhouser EM, Pulley L, Andrews JR, Osinski ED, Roseman JM. Longitudinal study of elbow and shoulder pain in youth baseball pitchers. Med Sci Sports Exerc. 2001 Nov;33(11):1803-10. doi: 10.1097/00005768-200111000-00002. PMID 11689728
- [Result] Lyman S, Fleisig GS, Andrews JR, Osinski ED. Effect of pitch type, pitch count, and pitching mechanics on risk of elbow and shoulder pain in youth baseball pitchers. Am J Sports Med. 2002 Jul-Aug;30(4):463-8. doi: 10.1177/03635465020300040201. PMID 12130397
- [Result] Dun S, Loftice J, Fleisig GS, Kingsley D, Andrews JR. A biomechanical comparison of youth baseball pitches: is the curveball potentially harmful? Am J Sports Med. 2008 Apr;36(4):686-92. doi: 10.1177/0363546507310074. Epub 2007 Nov 30. PMID 18055920
- [Result] Fleisig GS, Weber A, Hassell N, Andrews JR. Prevention of elbow injuries in youth baseball pitchers. Curr Sports Med Rep. 2009 Sep-Oct;8(5):250-4. doi: 10.1249/JSR.0b013e3181b7ee5f. PMID 19741352
- [Result] Nissen CW, Westwell M, Ounpuu S, Patel M, Solomito M, Tate J. A biomechanical comparison of the fastball and curveball in adolescent baseball pitchers. Am J Sports Med. 2009 Aug;37(8):1492-8. doi: 10.1177/0363546509333264. Epub 2009 May 15. PMID 19448049
- [Result] Dwelly PM, Tripp BL, Tripp PA, Eberman LE, Gorin S. Glenohumeral rotational range of motion in collegiate overhead-throwing athletes during an athletic season. J Athl Train. 2009 Nov-Dec;44(6):611-6. doi: 10.4085/1062-6050-44.6.611. PMID 19911087
- [Result] Bach HG, Goldberg BA. Posterior capsular contracture of the shoulder. J Am Acad Orthop Surg. 2006 May;14(5):265-77. doi: 10.5435/00124635-200605000-00002. PMID 16675620
- [Result] Grossman MG, Tibone JE, McGarry MH, Schneider DJ, Veneziani S, Lee TQ. A cadaveric model of the throwing shoulder: a possible etiology of superior labrum anterior-to-posterior lesions. J Bone Joint Surg Am. 2005 Apr;87(4):824-31. doi: 10.2106/JBJS.D.01972. PMID 15805213
- [Result] Trakis JE, McHugh MP, Caracciolo PA, Busciacco L, Mullaney M, Nicholas SJ. Muscle strength and range of motion in adolescent pitchers with throwing-related pain: implications for injury prevention. Am J Sports Med. 2008 Nov;36(11):2173-8. doi: 10.1177/0363546508319049. Epub 2008 Jul 2. PMID 18596197
- [Result] Nakamizo H, Nakamura Y, Nobuhara K, Yamamoto T. Loss of glenohumeral internal rotation in little league pitchers: a biomechanical study. J Shoulder Elbow Surg. 2008 Sep-Oct;17(5):795-801. doi: 10.1016/j.jse.2008.02.013. Epub 2008 Jun 20. PMID 18571440
- [Result] Olsen SJ 2nd, Fleisig GS, Dun S, Loftice J, Andrews JR. Risk factors for shoulder and elbow injuries in adolescent baseball pitchers. Am J Sports Med. 2006 Jun;34(6):905-12. doi: 10.1177/0363546505284188. Epub 2006 Feb 1. PMID 16452269
- [Result] Klingele KE, Kocher MS. Little league elbow: valgus overload injury in the paediatric athlete. Sports Med. 2002;32(15):1005-15. doi: 10.2165/00007256-200232150-00004. PMID 12457420
- [Result] Mair SD, Uhl TL, Robbe RG, Brindle KA. Physeal changes and range-of-motion differences in the dominant shoulders of skeletally immature baseball players. J Shoulder Elbow Surg. 2004 Sep-Oct;13(5):487-91. doi: 10.1016/j.jse.2004.02.008. PMID 15383802
- [Result] Reiss M, Reiss G. [Current aspects of handedness]. Wien Klin Wochenschr. 1999 Dec 23;111(24):1009-18. German. PMID 10677887
- See also: Youth baseball player reference site for help in reducing pain and injury from throwing — http://www.safethrow.com